CLINICAL TRIAL: NCT06949163
Title: Effect of Enteral Polymeric Formulas (Commercial and Homemade Formula) on Muscle Mass in Adults With Trauma Brain Injury
Brief Title: Effect of Enteral Formula (Commercial vs. Homemade) on Muscle Mass in Trauma Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital General "Dr. Miguel Silva" de Morelia (Other)
Responsible Party: Principal Investigator, KARINA AGUILAR GUTIERREZ, Karina Aguilar Gutiérrez, Hospital General "Dr. Miguel Silva" de Morelia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 666/02/23
Record Dates: First submitted 2025-04-22; First posted 2025-04-29 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: TBI Traumatic Brain Injury; Enteral Nutrition Therapy; Critical Illness
Keywords: Trauma brain injury; Enteral nutrition; Critically ill; Muscle Loss
MeSH Terms: conditions — Brain Injuries, Traumatic; Critical Illness; Muscular Atrophy

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Both the patient and the principal investigator will be blinded to the assigned formula.
  A hospital nutritionist will be responsible for the prescription and progression according to the proposed requirements and the tolerance of the assigned formula.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Homemade formula (Other): Patients receiving homemade formula made with natural food and will be administered according to the study protocol
  Interventions: Other: Homemade formula
- Commercial enteral formula (Other): Patients receiving commercial formula and will be administered according to the study protocol.
  Interventions: Dietary Supplement: Commercial formula

INTERVENTIONS:
Other: Homemade formula — Patients will receive enteral feeding with a polymeric formula made from blended natural foods (apple, chayote, cookie, chicken and olive oil), adjusted to meet their nutritional requirements (energy: 25 kcal/kg, protein: 1.3 g/kg).
  Other Names: blenderized tube feeding
  Arms: Homemade formula
Dietary Supplement: Commercial formula — Patients will receive enteral feeding with a commercial polymeric formula, adjusted to meet their nutritional requirements (energy: 25 kcal/kg, protein: 1.3 g/kg).
  Other Names: polymeric formula
  Arms: Commercial enteral formula

SUMMARY:
This randomized controlled clinical trial aims to determine whether there are differences in muscle mass (MM) in patients with traumatic brain injury who receive enteral nutrition based on polymeric formulas (homemade formula with blended natural foods versus commercial formulas).

DETAILED DESCRIPTION:
Patients admitted to the intensive care unit (ICU) with traumatic brain injury (TBI) lose MM, especially during the first ten days because it's used for organic, immune and tissue repair functions; the patients with moderate or severe TBI are frequently unable to eat food by themselves, so they receive enteral nutrition support (NS) with polymeric formulas. This support has been shown to attenuate muscle loss. Polymeric formulas can be industrially formulated or made with natural food, but there is no information available on their effect on MM using indicators such as femoral muscle thickness (femoral thickness, rectus femoris and vastus intermedius) by ultrasound (US) and phase angle (PhA) obtained by bioimpedance (BIA), as well as gastrointestinal tolerance (GIT).

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥ 18 years - 65 years
* Sex: Both sexes
* Moderate/severe TBI (Glasgow <13 points) admitted to the ICU
* Invasive mechanical ventilation >48 hours
* Candidates for enteral nutrition via nasogastric/orogastric tube

Exclusion Criteria:

* Pregnant women
* Patients with pacemakers
* Food allergies: egg, chicken, fish, nuts, or lactose intolerance
* Brain death
* Limb amputation or presence of external limb fixators

Elimination criteria:

* Withdrawal of consent
* Transfer to another healthcare institution.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2023-06-26 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
Femoral muscle (total femoral thickness, rectus femoris vastus intermedius) ultrasound | Change from baseline to end of study, an average of 10 days, with three measurements during follow-up (baseline, 5 days, and 10 days)
  Ultrasound-guided assessment of femoral muscle thickness. A certified intensivist physician accredited by the World Interactive Network Focused On Critical UltraSound, will perform duplicate measurements of muscle thicknesses (total femoral thickness, rectus femoris, and vastus intermedius) at the midpoint and one-third point of the distance between the superior border of the patella and the anterior superior iliac spine. The linear transducer will be positioned at a 90° angle to the thigh, without applying pressure (no compression). The average of the four measurements will then be calculated.

SECONDARY OUTCOMES:
Phase angle | Change from baseline to end of study, an average of 10 days, with three measurements during follow-up (baseline, 5 days, and 10 days)
  PhA was assessed using a multifrequency BIA analyzer with 8 limb electrodes, two electrodes per limb. Measurements were taken either two hours before or two hours after the formula infusion.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital General "Dr. Miguel Silva", Morelia, Michoacán, Mexico

IPD SHARING:
Plan to Share IPD: No
No, individual participant data (IPD) will not be shared with other researchers.
  The data collected are part of a small-scale, single-center study involving vulnerable patients in critical care. Due to concerns about patient confidentiality, limited sample size, and the absence of prior consent for data sharing beyond the original study scope, we have decided not to make IPD publicly available.

REFERENCES:
- [Background] Compher C, Bingham AL, McCall M, Patel J, Rice TW, Braunschweig C, McKeever L. Guidelines for the provision of nutrition support therapy in the adult critically ill patient: The American Society for Parenteral and Enteral Nutrition. JPEN J Parenter Enteral Nutr. 2022 Jan;46(1):12-41. doi: 10.1002/jpen.2267. Epub 2022 Jan 3. PMID 34784064
- [Background] Bechtold ML, Brown PM, Escuro A, Grenda B, Johnston T, Kozeniecki M, Limketkai BN, Nelson KK, Powers J, Ronan A, Schober N, Strang BJ, Swartz C, Turner J, Tweel L, Walker R, Epp L, Malone A; ASPEN Enteral Nutrition Committee. When is enteral nutrition indicated? JPEN J Parenter Enteral Nutr. 2022 Sep;46(7):1470-1496. doi: 10.1002/jpen.2364. Epub 2022 Jul 15. PMID 35838308
- [Background] Katari Y, Srinivasan R, Arvind P, Hiremathada S. Point-of-Care Ultrasound to Evaluate Thickness of Rectus Femoris, Vastus Intermedius Muscle, and Fat as an Indicator of Muscle and Fat Wasting in Critically Ill Patients in a Multidisciplinary Intensive Care Unit. Indian J Crit Care Med. 2018 Nov;22(11):781-788. doi: 10.4103/ijccm.IJCCM_394_18. PMID 30598564
- [Background] Nascimento TS, de Queiroz RS, Ramos ACC, Martinez BP, Da Silva E Silva CM, Gomes-Neto M. Ultrasound Protocols to Assess Skeletal and Diaphragmatic Muscle in People Who Are Critically Ill: A Systematic Review. Ultrasound Med Biol. 2021 Nov;47(11):3041-3067. doi: 10.1016/j.ultrasmedbio.2021.06.017. Epub 2021 Aug 18. PMID 34417065
- [Background] Epp L, Blackmer A, Church A, Ford I, Grenda B, Larimer C, Lewis-Ayalloore J, Malone A, Pataki L, Rempel G, Washington V; ASPEN Enteral Nutrition Committee. Blenderized tube feedings: Practice recommendations from the American Society for Parenteral and Enteral Nutrition. Nutr Clin Pract. 2023 Dec;38(6):1190-1219. doi: 10.1002/ncp.11055. Epub 2023 Oct 3. PMID 37787762
- [Background] Blenderized Feeding Options - The Sky's the Limit. Epp, L. June 2018, Practical Gastroenterology , pp. 30-39
- [Background] Voskuil C, Dudar M, Zhang Y, Carr J. Skeletal Muscle Ultrasonography and Muscle Fitness Relationships: Effects of Scanning Plane and Echogenicity Correction. Muscles. 2023 Mar 23;2(2):109-118. doi: 10.3390/muscles2020010. PMID 40757563
- [Background] Fazzini B, Markl T, Costas C, Blobner M, Schaller SJ, Prowle J, Puthucheary Z, Wackerhage H. The rate and assessment of muscle wasting during critical illness: a systematic review and meta-analysis. Crit Care. 2023 Jan 3;27(1):2. doi: 10.1186/s13054-022-04253-0. PMID 36597123
- [Background] Kalra S, Malik R, Singh G, Bhatia S, Al-Harrasi A, Mohan S, Albratty M, Albarrati A, Tambuwala MM. Pathogenesis and management of traumatic brain injury (TBI): role of neuroinflammation and anti-inflammatory drugs. Inflammopharmacology. 2022 Aug;30(4):1153-1166. doi: 10.1007/s10787-022-01017-8. Epub 2022 Jul 8. PMID 35802283
- [Background] Khellaf A, Khan DZ, Helmy A. Recent advances in traumatic brain injury. J Neurol. 2019 Nov;266(11):2878-2889. doi: 10.1007/s00415-019-09541-4. Epub 2019 Sep 28. PMID 31563989
- [Background] Bailes JE, Borlongan CV. Traumatic brain injury. CNS Neurosci Ther. 2020 Jun;26(6):593-594. doi: 10.1111/cns.13397. No abstract available. PMID 32452140